CLINICAL TRIAL: NCT05922436
Title: A Multicentre, Randomized, Double-blind, Parallel Design Phase III Study to Evaluate the Efficacy and Safety of Intravenous QLG2071 Versus Cleviprex® for Patients With Hypertensive Emergency and Sub-emergency
Brief Title: a Study Evaluating the Safety and Efficacy of Clevidipine for Patients Who With Hypertensive Emergency and Sub-emergency
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Pharmaceutical (Hainan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QLG2071-301
Record Dates: First submitted 2023-06-12; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Hypertensive Emergency
MeSH Terms: conditions — Hypertensive Crisis | interventions — clevidipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- QLG2071 (Experimental): QLG2071 25mg: 50ml
  Interventions: Drug: QLG2071
- Cleviprex® (Active Comparator): Cleviprex® 25mg: 50ml
  Interventions: Drug: Cleviprex®

INTERVENTIONS:
Drug: QLG2071 — intravenous injection
  Other Names: Clevidipine Butyrate Injectable Emulsion
  Arms: QLG2071
Drug: Cleviprex® — intravenous injection
  Other Names: Clevidipine Butyrate Injectable Emulsion
  Arms: Cleviprex®

SUMMARY:
A Multicentre, Randomized, Double-blind, Parallel Design Phase III Study to Evaluate the efficacy and safety of QLG2071 Versus Cleviprex® in the Treatment of Hypertensive Emergency and Sub-emergency

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, active-compared Phase III clinical study to evaluate the efficacy and safety of clevidipine butyrate injectable emulsion in the treatment of Hypertensive Emergency and Sub-emergency. The Cleviprex® will be chosen as the positive controlled medicine with the same usage of the test drug

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years-old and ≤75 years-old, regardless of gender;
2. Systolic blood pressure >180 mmHg and/or diastolic blood pressure >120 mmHg assessed on two successive occasions, 15 minutes apart at baseline；
3. Able to understand informed consent, participate in the experiment voluntarily and sign informed consent.

Exclusion Criteria:

1. Patients with known severe lipid metabolism disorders;
2. Patients with severe acute cardiovascular disease, such as confirmed or suspected severe aortic stenosis or aortic dissection, aortic syndrome, severe mitral stenosis, obstructive hypertrophic cardiomyopathy, acute myocardial infarction, and patients who have had an acute myocardial infarction within 1 month prior to signing the written informed consent;
3. Patients with acute ischemic/hemorrhagic stroke or cerebral hemorrhage within 1 month before signing the written informed consent;
4. Patients with known history of liver failure or cirrhosis and chronic kidney disease stage 5 requiring long-term regular dialysis treatment;
5. Patients with clear history of secondary hypertension;
6. Patients with other serious large organ damage or serious complications, it may threaten life;
7. Known intolerance to test drugs or calcium channel blockers; or who are allergic to soy, soy products, eggs, and egg products, or to experimental drug excipients;
8. Intravenous antihypertensive drugs have been used within 2 hours before the administration of test drugs;
9. Patients who cannot tolerate intravenous infusion therapy for at least 6 hours;
10. Pregnant and lactating women or patients who plan to have a family during the trial period;
11. Patients who have participated in other interventional clinical trials within 3 months prior to screening;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2024-05-24 (Estimated); Study Completion 2024-05-25 (Estimated)

PRIMARY OUTCOMES:
the percentage of patients who reach the target range (Systolic Blood Pressure decreased by ≥15% and ≤25% from baseline) within 30 minutes of administration | Within 30 minutes of the initiation of the infusion
  Proportion of patients who reach the target range within 30 minutes of administration

SECONDARY OUTCOMES:
The time for the first SBP fell within the target range (SBP decreased by ≥15% and ≤25% from baseline) within 30 minutes of administration | Within 30 minutes of the initiation of the infusion
  The time for the first SBP fell within the target range (SBP decreased by ≥15% and ≤25% from baseline) within 30 minutes of administration
Proportion of patients successfully converted to oral antihypertensive therapy within 6 hours of discontinuation | within 6 hours of discontinuation
  Proportion of patients successfully converted to oral antihypertensive therapy within 6 hours of discontinuation
Change in heart rate | within 30 minutes of administration
  Change of heart rate from baseline within 30 min of administration
Time to attainment of the 30-minute SBP target range | within 30 minutes of administration
  Time to attainment of the 30-minute SBP target range

OTHER OUTCOMES:
Incidence of adverse events (AEs) | Throughout the study period,up to 4 days
  Incidence of adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Yuguo Chen, Principal Investigator — Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: No